CLINICAL TRIAL: NCT00160134
Title: A Randomized, Placebo-Controlled, Double-Blind, Multi-Center, Parallel Group, Single Dose Study to Evaluate Cardiac Hemodynamics and Safety During Right Heart Catheterization of Three IV Doses of SLV320 in Subjects With Congestive Heart Failure Requiring Diuretic Treatment
Brief Title: Study to Evaluate Cardiac Hemodynamics and Safety of SLV320 in Subjects With Congestive Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S320.2.002; 2004-000442-21
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Congestive Heart Failure
Keywords: congestive heart failure, adenosine receptor blocker, cardiac hemodynamic
MeSH Terms: conditions — Heart Failure | interventions — SLV320 compound

INTERVENTIONS:
Drug: SLV320

SUMMARY:
The study is a randomized, placebo controlled, multi-center, single dose study to evaluate cardiac hemodynamics and safety of iv SLV320 in 110 subjects with congestive heart failure requiring diuretic treatment. Each subject will receive one dose of SLV320 or placebo or furosemide. The study consists of three visits (or study days when in-subjects are included). Ambulatory subjects will be in hospital for two nights and one day.

ELIGIBILITY:
Inclusion Criteria:

* history of chronic, symptomatic, mild to severe (NYHA Class II-IV) CHF for at least three months requiring treatment with diuretics and with documented systolic dysfunction
* on stable doses of their individually optimized medication regimen for at least one week prior to enrollment

Exclusion Criteria:

* required hospitalization (for cardiovascular disease) or adjustment of background medications for CHF
* orthostatic hypotension or symptomatic orthostasis
* sitting systolic or diastolic blood pressure < 90 mmHg
* 2nd or 3rd degree atrio-ventricular block or sick sinus syndrome
* heart rate of < 50 or > 110 bpm on the ECG
* transplanted heart
* heart failure due to primary valvular disease (unless surgically corrected), obstructive cardiomyopathy, pericardial disease, cor pulmonale or congenital heart disease
* hemodynamically significant left ventricular outflow tract obstruction

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (1):
- Site 1, Bad Nauheim, Germany

REFERENCES:
- [Derived] Mitrovic V, Seferovic P, Dodic S, Krotin M, Neskovic A, Dickstein K, de Voogd H, Bocker C, Ziegler D, Godes M, Nakov R, Essers H, Verboom C, Hocher B. Cardio-renal effects of the A1 adenosine receptor antagonist SLV320 in patients with heart failure. Circ Heart Fail. 2009 Nov;2(6):523-31. doi: 10.1161/CIRCHEARTFAILURE.108.798389. Epub 2009 Sep 24. PMID 19919976